CLINICAL TRIAL: NCT01051752
Title: Pharmacokinetics and Pharmacodynamics of Drugs for Nontuberculous Mycobacterial Diseases in Dutch Patients
Brief Title: PK and PD of Drugs for Nontuberculous Mycobacterial Diseases in Dutch Patients
Acronym: NTM
Status: Completed | Type: Observational
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: NL29420.091.09
Record Dates: First submitted 2010-01-18; First posted 2010-01-20 (Estimated); Last update posted 2012-05-22 (Estimated); Status verified 2012-05

CONDITIONS: Nontuberculous Mycobacterial Diseases
Keywords: Nontuberculous mycobacterial diseases; pharmacokinetics; pharmacodynamics

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples for pharmacokinetic analysis will be retained. Sputum samples for pharmacodynamic analysis will be retained.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- NTM infection: Patients with NTM infection are generally middle aged or higher aged, white males with COPD or bronchiectasis. They will be recruited from the outpatient clinics of University Centre for Chronic Diseases Dekkerswald, Tuberculosis Centre Beatrixoord or other outpatient clinics in The Netherlands. Both newly diagnosed and already treated patients with NTM disease will be recruited.

SUMMARY:
A prospective observational study in which pharmacokinetic and pharmacodynamic parameters are evaluated in a cohort of patients with NTM diseases.

DETAILED DESCRIPTION:
NTM are widely distributed in the environment and can especially be found in soil and water sources. These bacteria a very similar to tuberculosis bacteria. We are not that long aware that these bacteria can cause illness. Especially in patients with a chronic lung disease are sensitive to these bacteria and are susceptible to develop an infection. A lot of ambiguity consists about the best treatment of these infections. Up till now mainly the normal treatment for tuberculosis is used, however, the time period during which these medicines should be used and what dose should be used is mainly unknown.

To investigate whether the dose used at this moment is right a pharmacokinetic curve will be taken at steady-state.

ELIGIBILITY:
Inclusion Criteria:

* currently treated for NTM infection or recently diagnosed with NTM infection starting treatment at University Centre for Chronic Diseases Dekkerswald (Groesbeek), Centre for Revalidation Beatrixoord (Haren), or other outpatient clinics in The Netherlands.
* Diagnosis and treatment according to American Thoracic Society (ATS) criteria for NTM infections. Patients with pulmonary NTM infections (possible with extrapulmonary localizations as well) are eligible
* Treated with at least rifampicin and ethambutol and optionally with isoniazid, clarithromycin or azithromycin on a daily basis
* Age at least 18 years
* Patient has been using drugs for at least two weeks when steady state concentrations of the used drugs are expected
* Informed consent has been signed

Exclusion Criteria:

* The medical state of the patients does not allow inclusion according to the physician in attendance.
* The patients' clinical parameters urge immediate cessation of drugs.
* The patient is pregnant.
* Significant hepatic or renal dysfunction based on chemistry parameters (grade 1 according to an international adverse event grading system, see http:/ctep.cancer.gov) or symptomatic liver dysfunction (nausea and vomiting).
* Patients with cystic fibrosis, since these show deviating pharmacokinetics for many drugs.
* Patients with HIV infection, since these may show deviating pharmacokinetics for the drugs used in NTM disease.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with NTM infection are generally middle aged or higher aged, white males with COPD or bronchiectasis. They will be recruited from the outpatient clinics of University Centre for Chronic Diseases Dekkerswald, Tuberculosis Centre Beatrixoord or other outpatient clinics in The Netherlands. Both newly diagnosed and already treated patients with NTM disease will be recruited.
Sampling Method: Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2010-01; Primary Completion 2011-03 (Actual); Study Completion 2011-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic parameters of antimycobacterial drugs in NTM treatment | after at least 2 weeks of treatment

SECONDARY OUTCOMES:
Determinants of pharmacokinetic parameters | after at least 2 weeks of treatment
Assessment of MIC values and pharmacodynamic parameters for response | once a month starting after two weeks of treatment;last assessment at 6 months
Association of pharmacokinetic and pharmacodynamic parameters with treatment outcome and toxicity | entire study

CONTACTS AND LOCATIONS:
Overall Officials: Rob Aarnoutse, Pharm D PhD, Principal Investigator — Radboud University Medical Center; Jan- Willem Alffenaar, PharmD PhD, Principal Investigator — University Medical Center Groningen
Locations (2):
- Netherlands (2):
  - Radboud University Medical Centre Nijmegen, Nijmegen, Gelderland
  - University Medical Centre Groningen, Groningen, Provincie Groningen